CLINICAL TRIAL: NCT05766982
Title: Fish Skin Grafts With Platelet-rich Plasma Compared to Fish Skin Grafts for Chronic Wound Healing: Randomized, Prospective Trial
Brief Title: Kerecis Fish Skin Grafts With and Without Platelet Rich Plasma (PRP)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: St Elizabeth Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELD.001
Record Dates: First submitted 2023-03-02; First posted 2023-03-13 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Non-healing Wound
Keywords: xenograft; PRP; platelet rich plasma

STUDY DESIGN:
Intervention Model Description: This study will be a 1:1 randomized controlled trial with parallel group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Xenograft only (No Intervention): The Kerecis® xenograft (Kerecis® Omega3 MariGen) will be applied without the application of PRP.
- Xenograft and PRP (Experimental): The Kerecis® xenograft (Kerecis® Omega3 MariGen) will be applied with the application of PRP.
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Other: Platelet Rich Plasma — Platelet rich plasma will be applied to assess rate of wound healing.
  Arms: Xenograft and PRP

SUMMARY:
This prospective, randomized pilot study compares the use of a xenograft with PRP to a xenograft alone for chronic, nonhealing wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over the age of 18 years;
* The targeted wound is deemed a chronic, nonhealing wound after six weeks of treatment; - - Patient of Dr. Eldridge, Dr. Glenn, or Dr. Worley;
* Target wound size must be between 2 cm x 2 cm x 0.1 cm deep and 10 cm x 10 cm x 5 cm deep;
* Surgical candidate for standard of care Kerecis® xenograft surgery.

Exclusion Criteria:

* Patient with hemoglobin values less than 6.9 g/dL drawn at least 30 days prior to the Kerecis® xenograft surgery;
* Patient with a known allergy or other sensitivity to fish material;
* Patient is currently undergoing chemotherapy or radiation therapy;
* The targeted wound is of autoimmune origin; and Non-English-speaking patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Time to wound being deemed healed or 6 months | 6 months
  Assessed by time, surface area of wound, wound volume and relative surface size

SECONDARY OUTCOMES:
Wound quality of life | 6 months
  The Wound-QoL-14 questionnaire on quality of life with chronic wounds will be used to assess changes in score prior to initial application of xenograft or xenograft/PRP to time of wound healing or 6 months, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Elizabeth Healthcare Edgewood, Edgewood, Kentucky, United States